CLINICAL TRIAL: NCT05092334
Title: Effect of Proprioceptive Exercises on Pain and Function in Non-specific Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr//2043 Noshaba kanwal
Record Dates: First submitted 2021-09-13; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Neck Pain
Keywords: Neck disability index,; Numerical pain rating scale; Proprioceptive exercise
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive exercises (Experimental): Group A treated with proprioceptive exercises. proprioception exercises included.
  1. Head relocation it involve the practice of relocating head back to natural head posture and to predetermined positions in range first with eyes open using feedback from a laser attached to their head and then with closed all active movement of cervical flexion extension lateral flexion and rotations were used.
  2. Gaze stability oculomotor exercises commencing with eyes movement with the head stationary, progressing to movement of head with visual fixation on a target.
  3. Eye head coordination exercises, commenced with rotation of eyes and head to the same side in both right and left directions. Then progressed with both eyes and head move in opposite direction
  Interventions: Other: proprioceptive exercises
- Strengthening exercises (Experimental): Group B treated with strengthening exercises which are performed with prone and supine position by placing a towel under head, press towel for 5 seconds with 10-12 repetitions ,one set in a week for six weeks for cervical muscles
  Interventions: Other: Strengthening exercise

INTERVENTIONS:
Other: proprioceptive exercises — proprioception exercises included (a)Head relocation it involve the practice of relocating head back to natural head posture and to predetermined positions in range first with eyes open using feedback from a laser attached to their head and then with closed all active movement of cervical flexion extension lateral flexion and rotations were used.(b)Gaze stability oculomotor exercises commencing with eyes movement with the head stationary ,progressing to movement of head with visual fixation on a target. (c) Eye head coordination exercises, commenced with rotation of eyes and head to the same side in both right and left directions. Then progressed with both eyes and head move in opposite direction
  Arms: Proprioceptive exercises
Other: Strengthening exercise — strengthening exercises which are performed with prone and supine position by placing a towel under head, press towel for 5 seconds with 10-12 repetitions ,one set in a week for six weeks for cervical muscles
  Arms: Strengthening exercises

SUMMARY:
This study was conducted to see the effect of proprioceptive exercises on pain and function in Non-specific chronic neck pain.

Twenty participants with chronic Non-specific neck pain were enrolled in this study. During the final week of treatment, 14 patients were assessed at the end of the sixth treatment week. Participants were randomized into two groups treatment group and control group. Both groups were treated with conventional treatment which were strengthening exercises. Treatment group was also treated by proprioception exercises. For measurement of pain and disability NPRS and NDI scales were used. Exercise regime distributed in six weeks period one session per week exercise, 10-12 repetitions with 1-minute rest interval, lasted 45 minutes in both groups. pre-treatment and post-treatment measurements were taken.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific neck pain>3 months
* Postural neck pain

Exclusion Criteria:

* Vascular neoplasia
* Fibromyalgia
* Rheumatoid arthritis
* Radiculopathy
* Neuropathy
* Tumor
* Cervical fractures
* Vestibular problems
* Congenital disorder of cervical spine

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Numerical pain rating scale | 6 weeks
  11 point numeric scale ranges from 0 representing one pain extreme(no pain)to 10 representing the other pain extreme severity

SECONDARY OUTCOMES:
NECK DISABILITY INDEX | 6 weeks
  NDI is ten item questionnaire based on Oswestry low back pain that assess disability associated with neck pain and whiplash. There are four items that relate to symptoms(pain intensity ,headache, concentration ,sleeping)and six items that relate daily activities of life(lifting, work, driving, recreation, personal care, reading) 5-14 score :mild disability,15-24 score moderate disability,25-34 score severe disability,>35 complete disable

CONTACTS AND LOCATIONS:
Overall Officials: Qurat ul Ain, Mphil, Principal Investigator — Riphah International University
Locations (1):
- Qurat ul Ain, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coulter ID, Crawford C, Vernon H, Hurwitz EL, Khorsan R, Booth MS, Herman PM. Manipulation and Mobilization for Treating Chronic Nonspecific Neck Pain: A Systematic Review and Meta-Analysis for an Appropriateness Panel. Pain Physician. 2019 Mar;22(2):E55-E70. PMID 30921975